CLINICAL TRIAL: NCT01155193
Title: Prospective, Non-interventional Observation Study for the Use of Palivizumab in High-risk Children in Germany- SYNAGIS
Brief Title: Prospective Study for the Use of Palivizumab (Synagis®) in High-risk Children in Germany
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P10-410
Record Dates: First submitted 2010-03-02; First posted 2010-07-01 (Estimated); Results first posted 2018-10-29 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2017-07

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Children; Pre-term infants; Congenital heart disease; Infection; Respiratory syncytial virus; Bronchopulmonary dysplasia (BPD); Chronic lung disease (CLD)
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Heart Defects, Congenital; Infections; Bronchopulmonary Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Palivizumab: Participants were prescribed palivizumab (Synagis®) prophylaxis according to the German summary of product characteristics (SPC) for Synagis® to prevent serious disease due to RSV infection during the RSV season.

SUMMARY:
The SYNAGIS Registry was carried out in order to gather comprehensive real-world data on the use of palivizumab in children at high risk for serious respiratory syncytial virus (RSV) disease. This registry was designed as a post-marketing observational study, and conducted with the aim of collecting data on palivizumab administration, the risk factors for complicated RSV disease, frequency of hospitalizations, and drug adherence.

DETAILED DESCRIPTION:
Each participant included in this study was observed during his/her palivizumab prophylaxis during the prevailing RSV season. According to the requirements for non-interventional or observational studies, no diagnostic or monitoring procedures were applied to the participants included in the study other than those which would ordinarily be applied in the course of the individual therapeutic strategy. Only data which were part of routine medical care were collected.

Data collection was conducted initially in season 2002/2003 using paper-based case report forms (CRFs); beginning in season 2008/2009 a protected internet-based data entry platform was used. Both the paper-based CRFs and the electronic system were subject to changes during the whole time of the registry.

Data collection for registry seasons 2002/2003 - 2006/2007 was conducted by use of paper-based CRFs and hospitalization forms. Corresponding results were published in 2011 and are hence depicted together and reported here as a separate reporting group.

Registry seasons 2007/2008 and 2008/2009 were considered transitional years in the process of switching the type of data collection to an electronic CRF (eCRF) system. Although data collection of registry 2007/2008 was still paper-based, it was not included in the original publication and hence, results are reported separately. In season 2008/2009 the mode of data collection was switched from paper-based CRFs to an eCRF system, however, several physicians still used the paper-based CRFs for documentation. In order to use all documentations and lose as few data as possible, results for 2008/2009 are based on a combination of paper-based CRF and eCRF data. Hence, it was decided to keep the results for 08/09 separate from the depiction of the homogenous, eCRF-based results of the following seasons.

Data collection for registry 09/10 - 15/16 was implemented by an eCRF system. Corresponding results are therefore depicted together in one reporting group.

ELIGIBILITY:
Inclusion Criteria:

* Children born at 35 weeks of gestation or less and less than 6 months of age at the onset of the Respiratory syncytial virus season
* Children less than 2 years of age and requiring treatment for bronchopulmonary dysplasia within the last 6 months.
* Children less than 2 years of age and with hemodynamically significant congenital heart disease.

Exclusion Criteria:

* Children with known hypersensitivity to palivizumab or any component of the formulation, or other humanized monoclonal antibodies

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Primary care pediatricians from hospital outpatient facilities and neonatologists from inpatient facilities were invited to participate in this study and enrolled subjects into the registry at their discretion.
Sampling Method: Non-Probability Sample
Enrollment: 30804 (Actual)
Dates: Start 2002-09-01 (Actual); Primary Completion 2016-07-31 (Actual); Study Completion 2016-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Bloch, MD, Study Director — AbbVie Deutschland GmbH & Co. KG, Medical Department

REFERENCES:
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/drugInfo.cfm?id=41516

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pre-term infants and children under 24 months with high-risk for respiratory syncytial virus (RSV) were enrolled between September 01 and June 30 during each RSV season from 2002 to 2016. The registry was conducted in Germany.
Pre-assignment Details: Results were subdivided into four parts due to procedural changes including changes in the methods of study data reporting during the conduct of the study:
  * Registry 02/03 - 06/07
  * Registry 07/08
  * Registry 08/09
  * Registry 09/10 - 15/16
Groups:
- Palivizumab Registry 02/03 - 06/07: Participants were prescribed palivizumab (Synagis®) prophylaxis according to the German summary of product characteristics (SPC) for Synagis® to prevent serious disease due to RSV infection during the RSV season from 01 September 2002 until 30 June 2007.
- Palivizumab Registry 07/08: Participants were prescribed palivizumab (Synagis®) prophylaxis according to the German summary of product characteristics (SPC) for Synagis® to prevent serious disease due to RSV infection during the RSV season from 01 September 2007 to 30 June 2008.
- Palivizumab Registry 08/09: Participants were prescribed palivizumab (Synagis®) prophylaxis according to the German summary of product characteristics (SPC) for Synagis® to prevent serious disease due to RSV infection during the RSV season from 01 September 2008 to 30 June 2009.
- Palivizumab Registry 09/10 - 15/16: Participants were prescribed palivizumab (Synagis®) prophylaxis according to the German summary of product characteristics (SPC) for Synagis® to prevent serious disease due to RSV infection during the RSV season from 01 September 2009 to 30 June 2016.
Period: Overall Study
Arm/Group | Palivizumab Registry 02/03 - 06/07 | Palivizumab Registry 07/08 | Palivizumab Registry 08/09 | Palivizumab Registry 09/10 - 15/16
Started | 10924 | 3818 | 2260 | 13802
Completed | 10686 (Evaluable population (participants treated between 01 September and 01 May of the following year)) | 3805 (Evaluable population (participants treated between 01 September and 01 May of the following year)) | 2248 (Evaluable population (participants treated between 01 September and 01 May of the following year)) | 13711 (Evaluable population (participants treated between 01 September and 01 May of the following year))
Not Completed | 238 | 13 | 12 | 91

BASELINE CHARACTERISTICS:
Population: Evaluable population includes participants who received their first palivizumab injection between 01 September and 31 May of a given season, and who were younger than 2 years at start of immunoprophylaxis. For registry 09/10 - 15/16 only participants who received their first immunoprophylaxis in the corresponding season are included.
Groups:
- Palivizumab Registry 02/03 - 06/07: Participants were prescribed palivizumab (Synagis®) prophylaxis according to the German summary of product characteristics (SPC) for Synagis® to prevent serious disease due to RSV infection during the RSV season from 01 September 2002 to 30 June 2007.
- Total: Total of all reporting groups
Arm/Group | Palivizumab Registry 02/03 - 06/07 | Palivizumab Registry 07/08 | Palivizumab Registry 08/09 | Palivizumab Registry 09/10 - 15/16 | Total
Number analyzed (Participants) | 10686 | 3805 | 2248 | 12729 | 29468
Age, Customized [Count of Participants; unit: Participants] — Gestational age at birth is reported
  Participants
    < 29 weeks | 3582 | 1173 | 694 | 3514 | 8963
    29 to < 33 weeks | 3385 | 1161 | 705 | 4033 | 9284
    33 to ≤ 35 weeks | 1500 | 578 | 474 | 3237 | 5789
    > 35 weeks | 481 | 164 | 375 | 1945 | 2965
    Missing | 1738 | 729 | 0 | 0 | 2467
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 4901 | 1737 | 1019 | 5707 | 13364
  Male | 5716 | 2051 | 1229 | 7013 | 16009
  Missing | 69 | 17 | 0 | 9 | 95
Birth Weight [Count of Participants; unit: Participants]
  < 1000 g | 3283 | 1101 | 595 | 2946 | 7925
  1000 - 1499 g | 2782 | 965 | 538 | 3063 | 7348
  1500 - 1999 g | 1788 | 659 | 424 | 2590 | 5461
  ≥ 2000 g | 2595 | 995 | 691 | 4130 | 8411
  Missing | 238 | 85 | 0 | 0 | 323
Age at Start of Immunoprophylaxis [Mean (Standard Deviation); unit: months] — Population: Data are reported where available. Data are reported separately for different registry phases as no overall analysis was performed.
  months
    Registry 02/03 - 06/07: number analyzed (Participants) | 10059 | 0 | 0 | 0 | 10059
    Registry 02/03 - 06/07 | 5.2 (4.0) |  |  |  | 5.2 (4.0)
    Registry 07/08: number analyzed (Participants) | 0 | 3578 | 0 | 0 | 3578
    Registry 07/08 |  | 5.0 (4.0) |  |  | 5.0 (4.0)
    Registry 08/09: number analyzed (Participants) | 0 | 0 | 2248 | 0 | 2248
    Registry 08/09 |  |  | 5.9 (4.9) |  | 5.9 (4.9)
    Registry 09/10 - 15/16: number analyzed (Participants) | 0 | 0 | 0 | 12729 | 12729
    Registry 09/10 - 15/16 |  |  |  | 4.3 (3.6) | 4.3 (3.6)
Risk Factors for RSV Complications [Count of Participants; unit: Participants] — Population: Data are reported where available
  Participants
    Premature birth (< 29 weeks GA): number analyzed (Participants) | 8948 | 3076 | 2248 | 12729 | 27001
    Premature birth (< 29 weeks GA) | 3582 | 1173 | 694 | 3514 | 8963
    Premature birth (≤ 35 weeks GA): number analyzed (Participants) | 8948 | 3076 | 2248 | 12729 | 27001
    Premature birth (≤ 35 weeks GA) | 8467 | 2912 | 1873 | 10784 | 24036
    Multiple births: number analyzed (Participants) | 9752 | 3771 | 2141 | 12147 | 27811
    Multiple births | 2607 | 922 | 632 | 3793 | 7954
    Congenital heart disease: number analyzed (Participants) | 9588 | 3677 | 2248 | 12544 | 28057
    Congenital heart disease | 3001 | 1283 | 567 | 3430 | 8281
    Smoking in the family: number analyzed (Participants) | 8043 | 3031 | 2248 | 6332 | 19654
    Smoking in the family | 1422 | 482 | 400 | 2037 | 4341
    Chronic lung disease: number analyzed (Participants) | 9805 | 3501 | 2248 | 12422 | 27976
    Chronic lung disease | 4179 | 1330 | 584 | 2346 | 8439
    Immunodeficiency: number analyzed (Participants) | 8875 | 3428 | 2248 | 12271 | 26822
    Immunodeficiency | 430 | 167 | 30 | 171 | 798
    Attending daycare: number analyzed (Participants) | 9722 | 3745 | 2248 | 12389 | 28104
    Attending daycare | 240 | 109 | 74 | 361 | 784
    Other children (< 12 years) in household: number analyzed (Participants) | 9662 | 3728 | 2248 | 10767 | 26405
    Other children (< 12 years) in household | 4440 | 1682 | 1115 | 4899 | 12136
    Family history of asthma: number analyzed (Participants) | 7877 | 2956 | 2248 | 10589 | 23670
    Family history of asthma | 823 | 304 | NA — This risk factor was not assessed during this period | 1128 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Family history of allergic rhinitis: number analyzed (Participants) | 7819 | 2920 | 2248 | 12729 | 25716
    Family history of allergic rhinitis | 1234 | 450 | NA — This risk factor was not assessed during this period | NA — This risk factor was not assessed during this period | NA — Total not calculated because data are not available (NA) in one or more arms.
    Family history of allergic eczema: number analyzed (Participants) | 7751 | 2889 | 2248 | 12729 | 25617
    Family history of allergic eczema | 713 | 245 | NA — This risk factor was not assessed during this period | NA — This risk factor was not assessed during this period | NA — Total not calculated because data are not available (NA) in one or more arms.
    Family history of atopy: number analyzed (Participants) | 10686 | 3805 | 2248 | 10606 | 27345
    Family history of atopy | NA — This risk factor was not assessed during this period | NA — This risk factor was not assessed during this period | 346 | 2039 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Cyanotic heart defect: number analyzed (Participants) | 10686 | 3805 | 2248 | 12363 | 29102
    Cyanotic heart defect | NA — This risk factor was not assessed during this period | NA — This risk factor was not assessed during this period | 123 | 784 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Chronic lung disease therapy: number analyzed (Participants) | 10686 | 3805 | 2248 | 12291 | 29030
    Chronic lung disease therapy | NA — This risk factor was not assessed during this period | NA — This risk factor was not assessed during this period | 281 | 1803 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Treatment with oxygen at home: number analyzed (Participants) | 10686 | 3805 | 2248 | 12490 | 29229
    Treatment with oxygen at home | NA — This risk factor was not assessed during this period | NA — This risk factor was not assessed during this period | 133 | 763 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Neuromuscular impairment: number analyzed (Participants) | 10686 | 3805 | 2248 | 8435 | 25174
    Neuromuscular impairment | NA — This risk factor was not assessed during this period | NA — This risk factor was not assessed during this period | 120 | 786 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Down syndrome (Trisomy 21) | NA — This risk factor was not assessed during this period | NA — This risk factor was not assessed during this period | NA — This risk factor was not assessed during this period | 249 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Serious neurological disease: number analyzed (Participants) | 10686 | 3805 | 2248 | 8393 | 25132
    Serious neurological disease | NA — This risk factor was not assessed during this period | NA — This risk factor was not assessed during this period | NA — This risk factor was not assessed during this period | 428 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Low social status: number analyzed (Participants) | 10686 | 3805 | 2248 | 11915 | 28654
    Low social status | NA — This risk factor was not assessed during this period | NA — This risk factor was not assessed during this period | NA — This risk factor was not assessed during this period | 2258 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Crowded living conditions: number analyzed (Participants) | 10686 | 3805 | 2248 | 10575 | 27314
    Crowded living conditions | NA — This risk factor was not assessed during this period | NA — This risk factor was not assessed during this period | NA — This risk factor was not assessed during this period | 2592 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Exposition to air pollution: number analyzed (Participants) | 10686 | 3805 | 2248 | 10960 | 27699
    Exposition to air pollution | NA — This risk factor was not assessed during this period | NA — This risk factor was not assessed during this period | NA — This risk factor was not assessed during this period | 1710 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Breast feeding ≤ 2 months: number analyzed (Participants) | 10686 | 3805 | 2248 | 11417 | 28156
    Breast feeding ≤ 2 months | NA — This risk factor was not assessed during this period | NA — This risk factor was not assessed during this period | NA — This risk factor was not assessed during this period | 5794 | NA — Total not calculated because data are not available (NA) in one or more arms.
Immunoprophylaxis with Palivizumab Started in Hospital [Count of Participants; unit: Participants] — Population: Data are reported where available
  Participants
    number analyzed (Participants) | 10544 | 3745 | 1798 | 12729 | 28816
    (all) | 1645 | 519 | 313 | 3127 | 5604

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With RSV-associated Hospitalization
Time Frame: During RSV season (September to June) from 2002 to 2016
Population: Evaluable population with available hospitalization data
Measure: Number; unit: percentage of participants
Arm/Group | Palivizumab Registry 02/03 - 06/07 | Palivizumab Registry 07/08 | Palivizumab Registry 08/09 | Palivizumab Registry 09/10 - 15/16
Number analyzed (Participants) | 9833 | 3805 | 2248 | 12729
percentage of participants | 1.5 | 1.5 | 0.8 | 0.7

2. Secondary Outcome: Diagnosis Documented at Hospital Discharge in Registries 02/03 - 06/07 and 07/08
Description: Hospitalization due to RSV was documented on a separate hospitalization form. The data below represent the number of hospitalizations documented on forms; some participants may have had more than one hospitalization. Multiple entries for discharge diagnosis were possible.
Time Frame: During RSV season (September to June) from 2002 to 2008
Population: Participants in registries 02/03 - 06/07 and 07/08 who were hospitalized, and hospitalization was documented on paper case report forms.
Measure: Count of Units; unit: hospitalizations
Units Other Than Participants: hospitalizations
Arm/Group | Palivizumab Registry 02/03 - 06/07 | Palivizumab Registry 07/08
Number analyzed (Participants) | 324 | 107
Number analyzed (hospitalizations) | 334 | 121
hospitalizations
  Bronchiolitis | 67 | 18
  RSV-Bronchiolitis | 99 | 34
  Pneumonia (Viral pneumonia) | 26 | 12
  RSV-Pneumonia | 44 | 14
  RSV-Infection | 49 | 26
  Other | 134 | 70
  Any RSV diagnosis | 154 | 57

3. Secondary Outcome: Diagnosis Documented at Hospital Discharge in Registry 08/09 and 09/10 - 15/16
Description: In the season 2008/09, the eCRF system for data collection was introduced. Hospitalization due to RSV infection was documented on a separate hospitalization form in the electronic case report form (eCRF). Physicians were asked to specify a primary diagnosis at hospital discharge.
Time Frame: During RSV season (September to June) from 2008 to 2016
Population: Participants in registries 08/09 and 09/10 - 15/16 who were hospitalized, and hospitalization was documented on forms and with available diagnosis data (for registry 09/10 - 15/16)
Measure: Count of Units; unit: hospitalizations
Units Other Than Participants: hospitalizations
Groups:
- Registry 09/10 - 15/16 Hospitalization Associated With RSV: Participants who were prescribed palivizumab (Synagis®) prophylaxis according to the German SPC for Synagis® to prevent serious disease due to RSV infection during the RSV season from 01 September 2009 to 30 June 2016, and had a hospitalization associated with RSV infection.
- Registry 09/10 - 15/16 Hospitalizations Not RSV-Associated: Participants who were prescribed palivizumab (Synagis®) prophylaxis according to the German SPC for Synagis® to prevent serious disease due to RSV infection during the RSV season from 01 September 2009 to 30 June 2016, and had a hospitalization that was not associated with RSV infection.
Arm/Group | Palivizumab Registry 08/09 | Registry 09/10 - 15/16 Hospitalization Associated With RSV | Registry 09/10 - 15/16 Hospitalizations Not RSV-Associated
Number analyzed (Participants) | 79 | 87 | 269
Number analyzed (hospitalizations) | 90 | 85 | 220
hospitalizations
  Bronchitis | 24 | 24 | 115
  Bronchiolitis | 4 | 32 | 15
  Pneumonia (clinical diagnosis) | 7 | 9 | 27
  Pneumonia (confirmed by chest radiography) | 18 | 19 | 58
  Acute respiratory failure | 3 | 1 | 3
  Apnoea-bradycardia syndrome | 1 | 0 | 2
  Not specified | 33 | 0 | 0

4. Secondary Outcome: Presence of Complications During Hospitalization
Time Frame: During RSV season (September to June) from 2002 to 2016
Population: Evaluable population who were hospitalized and with available hospitalization complication data
Measure: Count of Units; unit: hospitalizations
Units Other Than Participants: hospitalizations
Groups:
- Registry 09/10 - 15/16 Hospitalization Associated With RSV: Participants who were prescribed palivizumab (Synagis®) prophylaxis according to the German SPC for Synagis® to prevent serious disease due to RSV infection during the RSV season from 01 September 2009 to 30 June 2016, and had a hospitalization that was associated with RSV infection.
Arm/Group | Palivizumab Registry 02/03 - 06/07 | Palivizumab Registry 07/08 | Palivizumab Registry 08/09 | Registry 09/10 - 15/16 Hospitalization Associated With RSV | Registry 09/10 - 15/16 Hospitalizations Not RSV-Associated
Number analyzed (Participants) | 324 | 107 | 79 | 87 | 269
Number analyzed (hospitalizations) | 334 | 121 | 90 | 92 | 356
hospitalizations
  Intensive care unit (ICU) admission: number analyzed (Participants) | 324 | 107 | 79 | 78 | 231
  Intensive care unit (ICU) admission: number analyzed (hospitalizations) | 334 | 121 | 90 | 83 | 308
  Intensive care unit (ICU) admission | 111 | 29 | 22 | 14 | 56
  Oxygen supplementation required: number analyzed (Participants) | 324 | 107 | 79 | 87 | 265
  Oxygen supplementation required: number analyzed (hospitalizations) | 334 | 121 | 90 | 92 | 352
  Oxygen supplementation required | 177 | 54 | 42 | 58 | 160
  Mechanical ventilation: number analyzed (Participants) | 324 | 107 | 79 | 72 | 213
  Mechanical ventilation: number analyzed (hospitalizations) | 334 | 121 | 90 | 75 | 286
  Mechanical ventilation | 44 | 11 | 8 | 6 | 34

5. Secondary Outcome: Parental Cooperation in Registries 02/03 - 06/07 and 07/08
Description: Cooperation of parents with the prophylaxis regimen was categorized as very good, good, moderate, bad or very bad.
Time Frame: During RSV season (September to June) from 2002 to 2008
Population: Evaluable population in registries 02/03 - 06/07 and 07/08
Measure: Count of Participants; unit: Participants
Arm/Group | Palivizumab Registry 02/03 - 06/07 | Palivizumab Registry 07/08
Number analyzed (Participants) | 10686 | 3805
Participants
  Very good/good | 9383 | 3340
  Moderate | 567 | 221
  Bad/very bad | 354 | 102
  Missing | 382 | 142

6. Secondary Outcome: Parental Cooperation for Registry 08/09 and 09/10 - 15/16
Description: Cooperation of parents with the prophylaxis regimen was evaluated per injection in registry 08/09 and 09/10 - 15/16. The categories for cooperation ratings were changed to good, satisfying, or bad:
  Good: all palivizumab doses could be administered as planned; Satisfying: a single palivizumab dose was missed by the parents; Bad: more than one palivizumab doses was missed by the parents.
Time Frame: During RSV season (September to June) from 2008 to 2016
Population: Evaluable population in in registries 08/09 and 09/10 - 15/16; for registry 09/10 - 15/16 only participants who received their first immunoprophylaxis in the corresponding season are included.
Measure: Count of Units; unit: Palivizumab injections
Units Other Than Participants: Palivizumab injections
Arm/Group | Palivizumab Registry 08/09 | Palivizumab Registry 09/10 - 15/16
Number analyzed (Participants) | 2248 | 12729
Number analyzed (Palivizumab injections) | 11039 | 63572
Palivizumab injections
  Good | 8175 | 51408
  Satisfying | 550 | 2985
  Bad | 143 | 575
  Missing | 2171 | 8604

7. Secondary Outcome: Mean Number of Palivizumab Injections
Description: The mean number of palivizumab injections per participant, per season.
Time Frame: During RSV season (September to June) from 2002 to 2016
Population: Evaluable population; for registry 09/10 - 15/16 only participants who received their first immunoprophylaxis in the corresponding season are included.
Measure: Mean (Standard Deviation); unit: palivizumab injections
Arm/Group | Palivizumab Registry 02/03 - 06/07 | Palivizumab Registry 07/08 | Palivizumab Registry 08/09 | Palivizumab Registry 09/10 - 15/16
Number analyzed (Participants) | 10686 | 3805 | 2248 | 12729
palivizumab injections | 4.7 (1.8) | 4.8 (1.9) | 4.9 (2.0) | 5.0 (2.0)

ADVERSE EVENTS:
Time Frame: During RSV season (June to September) from 2002 to 2016
Description: Evaluable population includes participants who received their first palivizumab injection between 01 September and 31 May of a given season, and who were younger than 2 years at start of immunoprophylaxis. For registry 09/10 - 15/16 only participants who received their first immunoprophylaxis in the corresponding season are included.
Groups:
- Palivizumab: Participants were prescribed palivizumab (Synagis®) prophylaxis according to the German summary of product characteristics (SPC) for Synagis® to prevent serious disease due to RSV infection during the RSV season (September to June) from 2002 to 2016.
Arm/Group | Palivizumab
Serious Adverse Events (participants affected / at risk) | 701/29468
Other Adverse Events (participants affected / at risk) | 34/29468
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palivizumab (N=29468)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 1
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 3
LEUKOPENIA (Blood and lymphatic system disorders) | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1
AORTIC VALVE STENOSIS (Cardiac disorders) | 1
BRADYCARDIA (Cardiac disorders) | 3
CARDIAC ARREST (Cardiac disorders) | 2
CARDIAC DISORDER (Cardiac disorders) | 2
CARDIAC FAILURE (Cardiac disorders) | 2
CARDIOPULMONARY FAILURE (Cardiac disorders) | 1
CARDIOVASCULAR INSUFFICIENCY (Cardiac disorders) | 1
CYANOSIS (Cardiac disorders) | 4
MYOCARDITIS (Cardiac disorders) | 1
RESTRICTIVE CARDIOMYOPATHY (Cardiac disorders) | 1
RIGHT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1
ATRIAL SEPTAL DEFECT (Congenital, familial and genetic disorders) | 1
CONGENITAL CENTRAL HYPOVENTILATION SYNDROME (Congenital, familial and genetic disorders) | 1
FALLOT'S TETRALOGY (Congenital, familial and genetic disorders) | 1
HEART DISEASE CONGENITAL (Congenital, familial and genetic disorders) | 2
HYPOPLASTIC LEFT HEART SYNDROME (Congenital, familial and genetic disorders) | 1
LISSENCEPHALY (Congenital, familial and genetic disorders) | 1
WOLF-HIRSCHHORN SYNDROME (Congenital, familial and genetic disorders) | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 1
DIAPHRAGMATIC HERNIA (Gastrointestinal disorders) | 1
DIARRHOEA (Gastrointestinal disorders) | 3
FLATULENCE (Gastrointestinal disorders) | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1
HAEMATOCHEZIA (Gastrointestinal disorders) | 1
INGUINAL HERNIA (Gastrointestinal disorders) | 1
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1
NECROTISING COLITIS (Gastrointestinal disorders) | 1
UMBILICAL HERNIA (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 4
ADVERSE DRUG REACTION (General disorders) | 6
ADVERSE EVENT (General disorders) | 2
CARDIAC DEATH (General disorders) | 1
DEATH (General disorders) | 12
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 12
HYPOTHERMIA (General disorders) | 1
MALAISE (General disorders) | 2
OEDEMA (General disorders) | 1
PYREXIA (General disorders) | 21
ANAPHYLACTIC REACTION (Immune system disorders) | 1
ADENOVIRAL UPPER RESPIRATORY INFECTION (Infections and infestations) | 1
BRONCHIOLITIS (Infections and infestations) | 31
BRONCHITIS (Infections and infestations) | 124
BRONCHITIS VIRAL (Infections and infestations) | 1
CELLULITIS (Infections and infestations) | 1
CONJUNCTIVITIS (Infections and infestations) | 3
DEVICE RELATED SEPSIS (Infections and infestations) | 1
EXANTHEMA SUBITUM (Infections and infestations) | 1
GASTROENTERITIS (Infections and infestations) | 7
GASTROENTERITIS NOROVIRUS (Infections and infestations) | 3
GASTROENTERITIS ROTAVIRUS (Infections and infestations) | 2
INFECTION (Infections and infestations) | 3
INFECTIVE PERICARDIAL EFFUSION (Infections and infestations) | 1
INFLUENZA (Infections and infestations) | 3
LARYNGOTRACHEITIS OBSTRUCTIVE (Infections and infestations) | 1
MYELITIS (Infections and infestations) | 1
NASOPHARYNGITIS (Infections and infestations) | 7
OSTEOMYELITIS (Infections and infestations) | 2
OTITIS MEDIA (Infections and infestations) | 3
PERTUSSIS (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 105
PNEUMONIA BACTERIAL (Infections and infestations) | 1
PNEUMONIA ESCHERICHIA (Infections and infestations) | 1
PNEUMONIA INFLUENZAL (Infections and infestations) | 1
PNEUMONIA RESPIRATORY SYNCYTIAL VIRAL (Infections and infestations) | 51
PNEUMONIA VIRAL (Infections and infestations) | 18
PSEUDOCROUP (Infections and infestations) | 4
RESPIRATORY SYNCYTIAL VIRUS BRONCHIOLITIS (Infections and infestations) | 85
RESPIRATORY SYNCYTIAL VIRUS BRONCHITIS (Infections and infestations) | 30
RESPIRATORY SYNCYTIAL VIRUS INFECTION (Infections and infestations) | 44
RESPIRATORY TRACT INFECTION (Infections and infestations) | 19
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 3
SEPSIS (Infections and infestations) | 1
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1
SUPERINFECTION BACTERIAL (Infections and infestations) | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 12
VIRAL INFECTION (Infections and infestations) | 5
INJECTION RELATED REACTION (Injury, poisoning and procedural complications) | 1
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1
ANTIMICROBIAL SUSCEPTIBILITY TEST RESISTANT (Investigations) | 1
BODY TEMPERATURE INCREASED (Investigations) | 1
BREATH SOUNDS ABNORMAL (Investigations) | 1
CATHETERISATION CARDIAC (Investigations) | 1
INFLUENZA VIRUS TEST POSITIVE (Investigations) | 1
OXYGEN SATURATION DECREASED (Investigations) | 7
RESPIRATORY SYNCYTIAL VIRUS TEST POSITIVE (Investigations) | 8
STAPHYLOCOCCUS TEST POSITIVE (Investigations) | 1
WEIGHT DECREASED (Investigations) | 2
DECREASED APPETITE (Metabolism and nutrition disorders) | 1
DEHYDRATION (Metabolism and nutrition disorders) | 3
DIET REFUSAL (Metabolism and nutrition disorders) | 6
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 4
FLUID INTAKE REDUCED (Metabolism and nutrition disorders) | 7
LACTOSE INTOLERANCE (Metabolism and nutrition disorders) | 1
MALNUTRITION (Metabolism and nutrition disorders) | 2
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 1
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
HAEMANGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
HISTIOCYTOSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 1
FEBRILE CONVULSION (Nervous system disorders) | 5
HYDROCEPHALUS (Nervous system disorders) | 3
INFANTILE SPASMS (Nervous system disorders) | 2
SEIZURE (Nervous system disorders) | 5
NEONATAL DISORDER (Pregnancy, puerperium and perinatal conditions) | 1
POOR WEIGHT GAIN NEONATAL (Pregnancy, puerperium and perinatal conditions) | 1
APATHY (Psychiatric disorders) | 1
RESTLESSNESS (Psychiatric disorders) | 2
RENAL DISORDER (Renal and urinary disorders) | 1
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 5
APNOEA (Respiratory, thoracic and mediastinal disorders) | 8
APPARENT LIFE THREATENING EVENT (Respiratory, thoracic and mediastinal disorders) | 1
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 2
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1
BRONCHIAL HYPERREACTIVITY (Respiratory, thoracic and mediastinal disorders) | 2
BRONCHIAL OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 1
BRONCHITIS CHRONIC (Respiratory, thoracic and mediastinal disorders) | 1
BRONCHOPULMONARY DYSPLASIA (Respiratory, thoracic and mediastinal disorders) | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 13
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 15
HYPERCAPNIA (Respiratory, thoracic and mediastinal disorders) | 2
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 2
INFANTILE APNOEA (Respiratory, thoracic and mediastinal disorders) | 3
IRREGULAR BREATHING (Respiratory, thoracic and mediastinal disorders) | 1
LARYNGEAL STENOSIS (Respiratory, thoracic and mediastinal disorders) | 1
NEONATAL HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1
OBSTRUCTIVE AIRWAYS DISORDER (Respiratory, thoracic and mediastinal disorders) | 3
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1
RALES (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY DISORDER (Respiratory, thoracic and mediastinal disorders) | 12
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 16
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1
TACHYPNOEA (Respiratory, thoracic and mediastinal disorders) | 2
ECZEMA INFANTILE (Skin and subcutaneous tissue disorders) | 1
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1
RASH (Skin and subcutaneous tissue disorders) | 1
CARDIAC OPERATION (Surgical and medical procedures) | 7
ELECTIVE PROCEDURE (Surgical and medical procedures) | 1
ENTEROSTOMY (Surgical and medical procedures) | 1
HERNIA REPAIR (Surgical and medical procedures) | 3
HOSPITALISATION (Surgical and medical procedures) | 114
ILEOSTOMY CLOSURE (Surgical and medical procedures) | 1
IMMUNISATION (Surgical and medical procedures) | 1
OXYGEN SUPPLEMENTATION (Surgical and medical procedures) | 9
PHARYNGEAL RECONSTRUCTION (Surgical and medical procedures) | 1
PLASTIC SURGERY OF THE LIPS AND MOUTH (Surgical and medical procedures) | 1
PULMONARY VALVE REPAIR (Surgical and medical procedures) | 1
AORTIC STENOSIS (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palivizumab (N=29468)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1
CARDIOVASCULAR DISORDER (Cardiac disorders) | 1
CYANOSIS (Cardiac disorders) | 1
HEART DISEASE CONGENITAL (Congenital, familial and genetic disorders) | 1
DIARRHOEA (Gastrointestinal disorders) | 3
VOMITING (Gastrointestinal disorders) | 1
ADMINISTRATION SITE REACTION (General disorders) | 1
ADVERSE DRUG REACTION (General disorders) | 2
ADVERSE EVENT (General disorders) | 1
DRUG INEFFECTIVE (General disorders) | 1
IRRITABILITY POSTVACCINAL (General disorders) | 1
PERIPHERAL SWELLING (General disorders) | 1
PYREXIA (General disorders) | 6
VACCINATION SITE REACTION (General disorders) | 1
BRONCHITIS (Infections and infestations) | 3
BRUCELLOSIS (Infections and infestations) | 1
INFECTION (Infections and infestations) | 1
RESPIRATORY SYNCYTIAL VIRUS BRONCHITIS (Infections and infestations) | 1
RESPIRATORY SYNCYTIAL VIRUS INFECTION (Infections and infestations) | 3
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1
VIRAL INFECTION (Infections and infestations) | 1
OVERDOSE (Injury, poisoning and procedural complications) | 1
VACCINATION COMPLICATION (Injury, poisoning and procedural complications) | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 1
DIET REFUSAL (Metabolism and nutrition disorders) | 1
FEEDING DISORDER (Metabolism and nutrition disorders) | 1
CONFUSIONAL STATE (Psychiatric disorders) | 1
PERSONALITY CHANGE (Psychiatric disorders) | 1
RESTLESSNESS (Psychiatric disorders) | 2
SCREAMING (Psychiatric disorders) | 1
BRONCHIAL OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1
RASH (Skin and subcutaneous tissue disorders) | 3
HOSPITALISATION (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.